CLINICAL TRIAL: NCT05727709
Title: Dynamic Changes of Torquetenovirus Load in Chinese Renal Transplant Recipients During Immunosuppressive Therapy: A Double-blind Multicenter Prospective Observational Cohort Study
Brief Title: Dynamic Changes of Torquetenovirus (TTV) Load in Chinese Renal Transplant Recipients
Acronym: TTV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Anapure BioScience (Unknown); Caibo MedTech (Unknown); SKM BioTech (Unknown)
Responsible Party: Principal Investigator, Gang Chen, Professor, Deputy director of Institute of OrganTransplantation, Tongji Hospital
Other Study IDs: CTTV study
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant Infection; Virus; Immunosuppression
Keywords: kidney transplantation; rejection; infection; donor specific antibodies; cell-free DNA; Torque Teno Virus; immuno-monitoring
MeSH Terms: conditions — Virus Diseases; Rejection, Psychology; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about dynamic changes of Torquetenovirus (TTV) load in Chinese renal transplant recipients. The main questions it aims to answer are:

* Is there correlation between TTV load and rejection?
* Is there correlation between TTV load and infection?
* Can changes in the TTV load of kidney transplant recipients predict rejection or infection?

Participants will:

* receive 13 follow-up visits within 1 year after kidney transplantation
* provide 2 ml of whole blood for TTV load testing and other related testing at each follow-up
* provide 10 ml of whole blood for dd-cfDNA testing at four follow-ups (1, 3, 6 and 12 months after transplantation)
* provide 1 ml of serum for donor-specific antibody testing at three follow-ups (1, 6 and 12 months after transplantation)

ELIGIBILITY:
Inclusion Criteria:

* Receiving ABO compatible renal allotransplantation from the initiation of the study to December 31, 2023
* Receiving tacrolimus /mycophenolate mofetil(or mycophenolic acid)/prednisone as maintenance immunosuppression after renal transplantation
* Receiving universal prophylaxis for CMV infection and PJP infection

Exclusion Criteria:

* Receiving combined liver-kidney, pancreas-kidney or heart-kidney transplantation
* Recipients with active hepatitis B or hepatitis C infection
* Recipients with anticipated irregular follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed as a national multi-center prospective observational double-blind cohort study. The main outcome measures are plasma Torque Teno Virus (TTV) load and the incidence of infection and acute rejection, which will be observed from day 1 before renal transplantation to 1 year after renal transplantation.The study population is renal transplant recipients. Double-blind refers to that both the medical staff in charge and the patients are blinded to the plasma TTV viral load at each follow-up visit, and this will be unblinded after the last follow-up visit of the last subject is completed.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Renal allograft biopsy and serum creatinine | From day0 to day365 after kidney transplantation
  Any biopsy-proven acute rejection (Banff criterea) and clinical diagnosed acute rejection

SECONDARY OUTCOMES:
Infection event | From day0 to day365 after kidney transplantation
  Any bacterial, fungal (including PJP), mycobacterial, or viral (including CMV viremia, EB viremia, BK Viremia, BK Viruria, etc.) infection requiring hospitalization or prolongation of hospitalization, or requiring intravenous antibiotics or therapeutic use of antiviral drugs, or requiring reduction of immunosuppressive drugs
donor-specific antibodies (DSA) | From day0 to day365 after kidney transplantation
  the development of de novo DSA or a 30% increase of MFI value in preformed DSA
donor derived cell-free DNA | From day0 to day365 after kidney transplantation
  An increase in absolute or percent donor derived-cell free DNA from 1 month post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, PhD, Principal Investigator — Tongji Hospital
Locations (5):
- China (5):
  - West China Hospital，Sichuan University, Chengdu
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Changhai Hospital affiliated to Naval Military Medical University, Shanghai
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact tongjihlunli@163.com

REFERENCES:
- [Background] Fishman JA. Opportunistic infections--coming to the limits of immunosuppression? Cold Spring Harb Perspect Med. 2013 Oct 1;3(10):a015669. doi: 10.1101/cshperspect.a015669. PMID 24086067
- [Background] Haas M, Loupy A, Lefaucheur C, Roufosse C, Glotz D, Seron D, Nankivell BJ, Halloran PF, Colvin RB, Akalin E, Alachkar N, Bagnasco S, Bouatou Y, Becker JU, Cornell LD, Duong van Huyen JP, Gibson IW, Kraus ES, Mannon RB, Naesens M, Nickeleit V, Nickerson P, Segev DL, Singh HK, Stegall M, Randhawa P, Racusen L, Solez K, Mengel M. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 2018 Feb;18(2):293-307. doi: 10.1111/ajt.14625. Epub 2018 Jan 21. PMID 29243394
- [Background] Ahlenstiel-Grunow T, Pape L. Novel ways to monitor immunosuppression in pediatric kidney transplant recipients-underlying concepts and emerging data. Mol Cell Pediatr. 2021 Jul 26;8(1):8. doi: 10.1186/s40348-021-00118-8. PMID 34309698
- [Background] De Vlaminck I, Khush KK, Strehl C, Kohli B, Luikart H, Neff NF, Okamoto J, Snyder TM, Cornfield DN, Nicolls MR, Weill D, Bernstein D, Valantine HA, Quake SR. Temporal response of the human virome to immunosuppression and antiviral therapy. Cell. 2013 Nov 21;155(5):1178-87. doi: 10.1016/j.cell.2013.10.034. PMID 24267896
- [Background] Maggi F, Focosi D, Statzu M, Bianco G, Costa C, Macera L, Spezia PG, Medici C, Albert E, Navarro D, Scagnolari C, Pistello M, Cavallo R, Antonelli G. Early Post-Transplant Torquetenovirus Viremia Predicts Cytomegalovirus Reactivations In Solid Organ Transplant Recipients. Sci Rep. 2018 Oct 19;8(1):15490. doi: 10.1038/s41598-018-33909-7. PMID 30341363
- [Background] Rezahosseini O, Drabe CH, Sorensen SS, Rasmussen A, Perch M, Ostrowski SR, Nielsen SD. Torque-Teno virus viral load as a potential endogenous marker of immune function in solid organ transplantation. Transplant Rev (Orlando). 2019 Jul;33(3):137-144. doi: 10.1016/j.trre.2019.03.004. Epub 2019 Apr 4. PMID 30981537
- [Background] Solis M, Velay A, Gantner P, Bausson J, Filipputtu A, Freitag R, Moulin B, Caillard S, Fafi-Kremer S. Torquetenovirus viremia for early prediction of graft rejection after kidney transplantation. J Infect. 2019 Jul;79(1):56-60. doi: 10.1016/j.jinf.2019.05.010. Epub 2019 May 14. PMID 31100359
- [Background] Focosi D, Maggi F. Torque teno virus monitoring in transplantation: The quest for standardization. Am J Transplant. 2019 May;19(5):1599-1601. doi: 10.1111/ajt.15194. Epub 2018 Dec 17. No abstract available. PMID 30468687
- [Background] Kulifaj D, Durgueil-Lariviere B, Meynier F, Munteanu E, Pichon N, Dube M, Joannes M, Essig M, Hantz S, Barranger C, Alain S. Development of a standardized real time PCR for Torque teno viruses (TTV) viral load detection and quantification: A new tool for immune monitoring. J Clin Virol. 2018 Aug;105:118-127. doi: 10.1016/j.jcv.2018.06.010. Epub 2018 Jun 11. PMID 29957546
- [Background] Fernandez-Ruiz M, Albert E, Gimenez E, Rodriguez-Goncer I, Andres A, Navarro D, Aguado JM. Early kinetics of Torque Teno virus DNA load and BK polyomavirus viremia after kidney transplantation. Transpl Infect Dis. 2020 Apr;22(2):e13240. doi: 10.1111/tid.13240. Epub 2020 Jan 9. No abstract available. PMID 31883425